CLINICAL TRIAL: NCT00940108
Title: A Phase II, Multicentre, Randomised, Observer-blind Study to Evaluate the Immunogenicity, Safety and Tolerability of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in Healthy Children Aged >= 6 Months to < 9 Years.
Brief Title: A Clinical Trial of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-CAL-09-60
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Influenza Caused by the Novel Influenza A (H1N1) Virus
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSL425 (15 mcg) (Experimental): 15 mcg of hemagglutinin antigen per dose. 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425
- CSL425 (30 mcg) (Experimental): 30 mcg of hemagglutinin antigen per dose. 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425

INTERVENTIONS:
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal-free
  Arms: CSL425 (15 mcg)
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal-free
  Arms: CSL425 (30 mcg)

SUMMARY:
The purpose of this study is to determine whether CSL425 is a safe and effective vaccine for eliciting an immune response to H1N1 influenza in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >= 6 months to < 9 years at the time of the first study vaccination.
* For children < 3 years of age at the time of first vaccination, born at or after 36 weeks of gestation.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza virus vaccine or allergy to eggs, chicken protein, thiomersal, neomycin, polymyxin, or any components of the Study Vaccine.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (5):
- Australia (5):
  - Study Site, Westmead, New South Wales
  - Study Site, Brisbane, Queensland
  - Study Site, North Adelaide, South Australia
  - Study Site, Carlton, Victoria
  - Study Site, Subiaco, Western Australia

REFERENCES:
- [Result] Nolan T, McVernon J, Skeljo M, Richmond P, Wadia U, Lambert S, Nissen M, Marshall H, Booy R, Heron L, Hartel G, Lai M, Basser R, Gittleson C, Greenberg M. Immunogenicity of a monovalent 2009 influenza A(H1N1) vaccine in infants and children: a randomized trial. JAMA. 2010 Jan 6;303(1):37-46. doi: 10.1001/jama.2009.1911. Epub 2009 Dec 21. PMID 20026597

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One randomized participant withdrew consent prior to vaccine administration and was not included in the participant flow data or in any analysis population.
Groups:
- CSL425 (15 mcg) Cohort A: Participants aged 6 months to less than 3 years received two doses of CSL425 (15 mcg of haemagglutinin antigen per 0.25 mL dose) by intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
- CSL425 (30 mcg) Cohort A: Participants aged 6 months to less than 3 years received two doses of CSL425 (30 mcg of haemagglutinin antigen per 0.5 mL dose) by intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
- CSL425 (15 mcg) Cohort B: Participants aged 3 years to less than 9 years received two doses of CSL425 (15 mcg of haemagglutinin antigen per 0.25 mL dose) by intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
- CSL425 (30 mcg) Cohort B: Participants aged 3 years to less than 9 years received two doses of CSL425 (30 mcg of haemagglutinin antigen per 0.5 mL dose) by intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
Period: Overall Study
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Started | 82 | 80 | 103 | 104
Completed | 77 | 71 | 100 | 99
Not Completed | 5 | 9 | 3 | 5
Not completed — Adverse Event | 2 | 4 | 0 | 2
Not completed — Withdrew Consent | 2 | 1 | 0 | 1
Not completed — Dose 2 contraindicated | 1 | 1 | 0 | 1
Not completed — Declined further vaccination | 0 | 1 | 3 | 0
Not completed — Refused - pyrexia after Dose 1 | 0 | 1 | 0 | 0
Not completed — Viral illness after Dose 1 | 0 | 1 | 0 | 0
Not completed — Diagnosed with H1N1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B | Total
Number analyzed (Participants) | 82 | 80 | 103 | 104 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.68 (0.67) | 1.73 (0.74) | 5.78 (1.69) | 5.66 (1.74) | 3.96 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 53 | 49 | 184
  Male | 41 | 39 | 50 | 55 | 185

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titre Seroconversion Rate After the First Vaccination
Description: HI antibody titre seroconversion was defined as participants with a pre-vaccination titre of less than 1:10 achieving a post-vaccination HI antibody titre of 1:40 or more; or participants with a pre-vaccination HI titre of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titre.
Time Frame: Before and 21 days after the first vaccination
Population: The Evaluable Population (for the first vaccination) comprised all randomised participants who received the first study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 76 | 73 | 98 | 99
percentage of participants | 88.2 [78.7 to 94.4] | 97.3 [90.5 to 99.7] | 85.7 [77.2 to 92.0] | 91.9 [84.7 to 96.4]

2. Primary Outcome: HI Antibody Titre Seroconversion Rate After the Second Vaccination
Description: as for outcome 1
Time Frame: Before and 21 days after the second vaccination
Population: The Evaluable Population (for the second vaccination) comprised all randomised participants who received the second study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 64 | 69 | 95 | 96
percentage of participants | 96.9 [89.2 to 99.6] | 98.6 [92.2 to 100.0] | 97.9 [92.6 to 99.7] | 96.9 [91.1 to 99.4]

3. Primary Outcome: Geometric Mean Fold Increase (GMFI) in the HI Antibody Titre After the First Vaccination
Description: GMFI in HI antibody titre was defined as the geometric mean of the fold increase in the post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Before and 21 days after the first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 76 | 73 | 98 | 99
geometric mean fold increase | 13.95 [11.39 to 17.09] | 22.17 [17.87 to 27.49] | 13.25 [10.84 to 16.19] | 15.93 [12.87 to 19.71]

4. Primary Outcome: GMFI in the HI Antibody Titre After the Second Vaccination
Description: as for outcome 3
Time Frame: Before and 21 days after the second vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 64 | 69 | 95 | 96
geometric mean fold increase | 57.64 [42.87 to 77.50] | 72.93 [56.10 to 94.80] | 37.48 [28.33 to 49.58] | 37.06 [28.77 to 47.75]

5. Primary Outcome: Percentage of Participants Achieving a HI Antibody Titre of 1:40 or More After the First Vaccination
Time Frame: 21 days after the first vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 76 | 73 | 98 | 99
percentage of participants | 92.1 [83.6 to 97.0] | 100.0 [95.1 to 100.0] | 92.9 [85.8 to 97.1] | 96.0 [90.0 to 98.9]

6. Primary Outcome: Percentage of Participants Achieving a HI Antibody Titre of 1:40 or More After the Second Vaccination
Time Frame: 21 days after the second vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 64 | 69 | 95 | 96
percentage of participants | 100.0 [94.4 to 100.0] | 100.0 [94.8 to 100.0] | 100.0 [96.2 to 100.0] | 100.0 [96.2 to 100.0]

7. Secondary Outcome: Frequency and Intensity of Solicited Adverse Events (AEs) After the First or Second Vaccination
Description: Solicited AEs included AEs that were specifically sought for. Grade 3 solicited AE definitions: Cried when limb was moved/spontaneously painful (Cohort A) or prevented normal daily activities (Cohort B) for injection site pain; Size > 100 mm for injection site redness and induration/swelling; Temperature > 103.1°F (39.5°C) for fevers; Prevented normal daily activities or required medical intervention for all other systemic AEs.
Time Frame: During the 7 days after each vaccination
Population: The Safety Population comprised all participants who received at least one dose of the vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 82 | 80 | 103 | 104
percentage of participants
  Any solicited local AE | 69.5 | 63.8 | 68.0 | 71.2
  Any pain at injection site | 48.8 | 43.8 | 59.2 | 64.4
  Grade 3 pain at injection site | 1.2 | 1.3 | 0 | 1.0
  Any redness at injection site | 53.7 | 38.8 | 37.9 | 37.5
  Grade 3 redness at injection site | 0 | 1.3 | 2.9 | 2.9
  Any swelling/induration at injection site | 30.5 | 32.5 | 25.2 | 26.9
  Grade 3 swelling/induration at injection site | 0 | 2.5 | 0 | 4.8
  Any solicited systemic AE | 79.3 | 93.8 | 54.4 | 61.5
  Any nausea/vomiting | 13.4 | 30.0 | 15.5 | 20.2
  Grade 3 nausea/vomiting | 1.2 | 1.3 | 0 | 1.0
  Any diarrhoea | 26.8 | 32.5 | 12.6 | 12.5
  Grade 3 diarrhoea | 1.2 | 0 | 0 | 0
  Any loss of appetite | 40.2 | 50.0 | NA — Not solicited for in Cohort B | NA — Not solicited for in Cohort B
  Grade 3 loss of appetite | 1.2 | 0 | NA — Not solicited for in Cohort B | NA — Not solicited for in Cohort B
  Any irritability | 63.4 | 72.5 | NA — Not solicited for in Cohort B | NA — Not solicited for in Cohort B
  Grade 3 irritability | 2.4 | 1.3 | NA — Not solicited for in Cohort B | NA — Not solicited for in Cohort B
  Any fever | 50.0 | 71.3 | 20.4 | 29.8
  Grade 3 fever | 1.2 | 8.8 | 0 | 2.9
  Any headache | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 27.2 | 23.1
  Grade 3 headache | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 0 | 1.0
  Any muscle ache | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 15.5 | 22.1
  Grade 3 muscle ache | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 0 | 1.0
  Any malaise | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 19.4 | 26.9
  Grade 3 malaise | NA — Not solicited for in Cohort A | NA — Not solicited for in Cohort A | 0 | 1.9

8. Secondary Outcome: Duration of Solicited AEs After the First Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: During the 7 days after the first vaccination and up to Day 20 after the first vaccination if AE is ongoing at Day 7.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 82 | 80 | 103 | 104
days
  Pain at injection site | 1.48 (0.677) | 1.52 (0.823) | 1.91 (1.221) | 1.80 (1.016)
  Redness at injection site | 2.08 (1.382) | 2.23 (1.602) | 2.26 (1.347) | 2.00 (1.134)
  Swelling/induration at injection site | 1.88 (0.957) | 1.64 (0.745) | 1.60 (0.737) | 2.04 (1.136)
  Nausea/vomiting | 1.33 (0.500) | 1.05 (0.213) | 1.18 (0.405) | 1.53 (1.837)
  Diarrhoea | 1.67 (1.328) | 1.55 (0.945) | 1.11 (0.333) | 1.17 (0.577)
  Loss of appetite | 2.32 (1.906) | 1.97 (1.447) | NA (NA) — Not solicited for in Cohort B | NA (NA) — Not solicited for in Cohort B
  Irritability | 1.78 (1.560) | 1.73 (1.574) | NA (NA) — Not solicited for in Cohort B | NA (NA) — Not solicited for in Cohort B
  Fever | 1.77 (1.547) | 1.52 (1.079) | 1.40 (0.737) | 1.54 (1.319)
  Headache | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 2.04 (2.911) | 1.63 (1.149)
  Muscle ache | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 1.45 (0.688) | 1.86 (2.175)
  Malaise | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 1.60 (0.910) | 1.69 (1.966)

9. Secondary Outcome: Duration of Solicited AEs After the Second Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: During the 7 days after the second vaccination and up to Day 20 after the second vaccination if AE was ongoing at Day 7.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 77 | 71 | 100 | 99
days
  Pain at injection site | 1.67 (0.966) | 1.64 (1.002) | 1.90 (1.179) | 1.80 (1.040)
  Redness at injection site | 1.69 (1.004) | 2.14 (1.037) | 1.92 (1.055) | 1.70 (0.822)
  Swelling/induration at injection site | 1.74 (0.872) | 2.32 (1.108) | 2.24 (1.348) | 2.27 (1.751)
  Nausea/vomiting | 5.00 (8.832) | 1.00 (0.000) | 1.43 (0.787) | 1.11 (0.333)
  Diarrhoea | 3.40 (3.777) | 1.25 (0.452) | 1.40 (0.894) | 2.00 (1.000)
  Loss of appetite | 3.15 (4.475) | 1.73 (0.883) | NA (NA) — Not solicited for in Cohort B | NA (NA) — Not solicited for in Cohort B
  Irritability | 2.57 (2.410) | 2.10 (1.533) | NA (NA) — Not solicited for in Cohort B | NA (NA) — Not solicited for in Cohort B
  Fever | 2.14 (3.005) | 1.63 (1.165) | 1.54 (0.877) | 1.67 (1.414)
  Headache | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 1.33 (0.686) | 1.73 (2.412)
  Muscle ache | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 1.60 (0.516) | 1.29 (0.756)
  Malaise | NA (NA) — Not solicited for in Cohort A | NA (NA) — Not solicited for in Cohort A | 1.20 (0.422) | 2.00 (1.826)

10. Secondary Outcome: Incidence of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and New Onset of Chronic Illnesses (NOCIs)
Description: An AESI was defined as an AE for which the association with seasonal influenza vaccine was unclear. A NOCI was defined as the diagnosis of a new medical condition that was chronic in nature, including those potentially controllable by medication (eg, diabetes, asthma).
Time Frame: Up to 180 days after the last vaccination
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 82 | 80 | 103 | 104
percentage of participants
  At least one SAE | 4.9 | 1.3 | 1.0 | 1.0
  Related SAE | 0 | 0 | 0 | 1.0
  At least one AESI | 2.4 | 1.3 | 0 | 0
  Related AESI | 0 | 0 | 0 | 0
  At least one NOCI | 1.2 | 3.8 | 1.9 | 0
  Related NOCI | 0 | 0 | 0 | 0

11. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events After the First or Second Vaccination
Description: Unsolicited AEs included AEs other than those specifically sought for. Grade 1 unsolicited AE definition: Easily tolerated and did not interfere with normal daily activities. Grade 2 unsolicited AE definition: Some interference with normal daily activities. Grade 3 unsolicited AE definition: Prevented normal daily activities.
Time Frame: During the 21 days after each vaccination; up to 180 days after the last vaccination for SAEs, AESIs, and NOCIs
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Number analyzed (Participants) | 82 | 80 | 103 | 104
percentage of participants
  At least one unsolicited AE | 78.0 | 82.5 | 67.0 | 76.0
  Grade 1 unsolicited AE | 26.8 | 33.8 | 27.2 | 37.5
  Grade 2 unsolicited AE | 41.5 | 41.3 | 37.9 | 26.9
  Grade 3 unsolicited AE | 9.8 | 7.5 | 1.9 | 11.5

ADVERSE EVENTS:
Time Frame: For SAEs: up to 180 days after the last vaccination. For Other AEs: solicited AEs: during the 7 days after each vaccination; unsolicited AEs: during the 21 days after each vaccination; up to 180 days after the last vaccination for AESIs and NOCIs.
Description: Unsolicited AEs presented in the organ system "General disorders" with a footnote of "MedDRA V13.0", were collected under the MedDRA System Organ Class (SOC) 'General disorders and administration site conditions'. Solicited AEs are presented in the organ system "General disorders" and were not collected under the MedDRA SOC.
Arm/Group | CSL425 (15 mcg) Cohort A | CSL425 (30 mcg) Cohort A | CSL425 (15 mcg) Cohort B | CSL425 (30 mcg) Cohort B
Serious Adverse Events (participants affected / at risk) | 4/82 | 1/80 | 1/103 | 1/104
Other Adverse Events (participants affected / at risk) | 81/82 | 78/80 | 91/103 | 96/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL425 (15 mcg) Cohort A (N=82) | CSL425 (30 mcg) Cohort A (N=80) | CSL425 (15 mcg) Cohort B (N=103) | CSL425 (30 mcg) Cohort B (N=104)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CSL425 (15 mcg) Cohort A (N=82) | CSL425 (30 mcg) Cohort A (N=80) | CSL425 (15 mcg) Cohort B (N=103) | CSL425 (30 mcg) Cohort B (N=104)
Upper respiratory tract infection (Infections and infestations) | 22 (28) | 28 (31) | 22 (26) | 24 (26)
Viral infection (Infections and infestations) | 4 (4) | 0 (0) | 3 (4) | 9 (9)
Croup infectious (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Otitis media (Infections and infestations) | 4 (5) | 1 (1) | 3 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 8 (8) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12) | 13 (13) | 11 (12)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 17 (17) | 4 (4) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (6) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Influenza-like illness (General disorders) | 12 (14) | 10 (10) | 7 (8) | 9 (9)
Pyrexia (General disorders) | 10 (10) | 4 (4) | 3 (4) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 6 (6) | 4 (5) | 7 (7)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3) | 6 (8)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 0 (0) | 4 (5)
Hand-foot-and-mouth disease (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (4) | 2 (2)
Teething (Gastrointestinal disorders) | 14 (18) | 12 (19) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 0 (0) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain at Injection Site (General disorders) | 40 (52) | 35 (47) | 61 (96) | 67 (105)
Redness at Injection Site (General disorders) | 44 (66) | 31 (44) | 39 (53) | 39 (52)
Swelling/Induration at Injection Site (General disorders) | 25 (35) | 26 (33) | 26 (32) | 28 (40)
Nausea/Vomiting (General disorders) | 11 (15) | 24 (26) | 16 (18) | 21 (28)
Diarrhoea (General disorders) | 22 (28) | 26 (32) | 13 (14) | 13 (15)
Loss of Appetite (General disorders) | 33 (48) | 40 (55) | 0/0 (0) | 0/0 (0) — Not solicited for in Cohort B.
Irritability (General disorders) | 52 (92) | 58 (99) | 0/0 (0) | 0/0 (0) — Not solicited for in Cohort B.
Fever (General disorders) | 41 (51) | 57 (75) | 21 (28) | 31 (37)
Headache (General disorders) | 0/0 (0) | 0/0 (0) | 28 (42) | 24 (38) — Not solicited for in Cohort A.
Muscle Ache (Myalgia) (General disorders) | 0/0 (0) | 0/0 (0) | 16 (21) | 23 (28) — Not solicited for in Cohort A.
Malaise (General disorders) | 0/0 (0) | 0/0 (0) | 20 (25) | 28 (39) — Not solicited for in Cohort A.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.